CLINICAL TRIAL: NCT00171444
Title: A 8-week Comparison, in a General Practice Setting, Between Two Treatment Strategies With Valsartan and Valsartan/HCTZ Aiming at Normalizing de Novo Hypertensive Patients Who Are Not Adequately Controlled With Their Monotherapy or Biotherapy Treatment or Experiencing Unacceptable Side-effects, According to Their Baseline Blood Pressure
Brief Title: Comparison of Two Treatment Strategies in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CVAH631DFR06
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: hypertension,; valsartan+hydrochlorothiazide
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Medical education

SUMMARY:
The purpose of the study is to determine whether a specific training of General Practitioners (Family Physicians) regarding the new official guidelines for the treatment of hypertension results in a higher control of high Blood pressure in their patient population.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female patients >18 years of age

  * Hypertension defined by MSDBP ≥ 90 and /or MSSBP ≥ 140 mmHg for untreated patients, patients on diet and exercise, patients on current anti-hypertensive monotherapy or bitherapy treatment who remain uncontrolled or patients experiencing unacceptable side-effects,

Exclusion Criteria:

* • Severe hypertension, secondary hypertension, type 1 diabetes mellitus

  * History of congestive heart failure, unstable coronary insufficiency, life threatening arrhythmia, significant valvular disease, second or third degree heart block etc.
  * Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 4445 (Actual)
Dates: Start 2004-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure less than 140/90 mmHg in non-diabetic patients, or less than 130/80 mmHg in patients with diabetes or kidney disease, after 8 weeks

SECONDARY OUTCOMES:
Change from baseline systolic blood pressure after 8 weeks
Change from baseline diastolic blood pressure after 8 weeks
Diastolic blood pressure less than 90 mmHg or reduction in diastolic blood pressure greater than 10 mmHg
Systolic blood pressure less than 140 mmHg or reduction in diastolic blood pressure greater than 15 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novatis Pharmaceuticals